CLINICAL TRIAL: NCT05185531
Title: A Phase Ib Study of Neoadjuvant Tislelizumab With Stereotactic Body Radiotherapy in Patients With Resectable Hepatocellular Carcinoma
Brief Title: A Study of Neoadjuvant Tislelizumab With SBRT in Patients With Resectable Hepatocellular Carcinoma
Acronym: Notable-HCC
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Principal Investigator, Lei ZHAO, Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Notable-HCC
Record Dates: First submitted 2021-12-19; First posted 2022-01-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: neoadjuvant; PD-1; stereotactic body radiotherapy, SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant (Experimental): PD-1(Tislelizumab) plus stereotactic body radiotherapy
  Interventions: Combination Product: PD-1 plus stereotactic body radiotherapy

INTERVENTIONS:
Combination Product: PD-1 plus stereotactic body radiotherapy — neoadjuvant PD-1(Tislelizumab) plus stereotactic body radiotherapy (8 Gy × 3 fractions) in resectable HCC

SUMMARY:
Notable-HCC is a phase Ib study of neoadjuvant stereotactic body radiotherapy (SBRT) plus Programmed cell death-1 (PD-1, Tislelizumab, BeiGene) prior to hepatic resection in patients with resectable HCC.

DETAILED DESCRIPTION:
A baseline core tumor biopsy and peripheral venous blood will be collected from eligible participants at screening, and sample tumor tissue from the surgical specimen and PBMC (peripheral blood mononuclear cell) will be snap-frozen and stored for the future relevant studies.

Eligible patients will receive SBRT (8 Gy × 3 fractions, every other day) on day 1, day 3 and day 5; the first dose of Tislelizumab will be administrated concurrently on day 1, then the second on day 22 (the first day of week 4, ± 3 days). Then on day 50 (the first day of week 8, ± 7 days), curative liver resection of HCC will be scheduled.

Patients will be reviewed following completion of SBRT and tislelizumab treatment (Follow-up visit 1; FU1) prior to surgery.

Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) and HCC-Specific mRECIST criteria will be used to determine patient response to treatment, including CR (complete response), PR (partial response) and ORR (objective response rate). PBMC will be collected again and stored.

Hepatic resection will be performed as per standard of care. The safety FU2 will be conducted after the first dose of the post-resection tislelizumab. All AEs that occur prior to the visit will be recorded. Participants with on-going AEs at the visit will be followed up by principal investigator (PI) or delegate until resolution or stabilization of the event. Following FU2, participants will be assessed every 3 months (±7 days) thereafter to collect information regarding disease status and survival. Long-term follow-up will continue, for each patient, for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for the trial.
2. Aged ≥18 years
3. Willing to provide tissue from an excisional biopsy of a tumor lesion
4. Confirmed diagnosis of HCC. The diagnosis can be established radiographically by the criteria of the American Association for the Study of the Liver (AASLD), or by histologic diagnosis from the core biopsy.
5. Have measurable disease by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI) defined by RECIST (Response Evaluation Criteria In Solid Tumours) 1.1 criteria and HCC specific mRECIST (modified RECIST).
6. Medically fit to undergo surgery as determined by the treating medical and surgical oncology team
7. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1
8. Adequate organ and marrow function as defined below:

1) leukocytes ≥3,000/mcL 2) absolute neutrophil count ≥1,500/mcL 3) platelets ≥100,000/mcL 4) total bilirubin ≤ 2 × institutional upper limit of normal (ULN) 5) AST (aspartate aminotransferase)/ALT(alanine aminotransferase) ≤ 3 × institutional ULN 6) creatinine ≤ 1.5 × institutional ULN OR 7) estimated glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 (according to the Cockcroft-Gault formula) 9. Overall Child-Pugh class A 10. Documented virology status of hepatitis, as confirmed by screening tests for HBV (hepatitis B virus) and HCV (hepatitis C virus)

1. For patients with active HBV: HBV DNA <2000 IU/mL during screening, and have initiated anti-HBV treatment at least 14 days prior to SBRT and willingness to continue anti-HBV treatment during the study (per local standard of care; e.g., entecavir).
2. Patients with HCV, either with resolved infection (as evidenced by detectable antibody and negative viral load) or chronic infection (as evidenced by detectable HCV RNA), are eligible.

11. Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

12. Female patient of childbearing potential should have a negative serum pregnancy test within 24 h of her first dose of IMP (Investigational Medicinal Product) 13. Women of childbearing potential must be willing to use a highly effective method of contraception for the course of the study through 5 months after the last dose of IMP. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

14. Sexually active males must agree to use an adequate method of contraception starting with the first dose of IMP through 7 months after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.

Exclusion Criteria:

1. Extrahepatic metastasis
2. Prior systemic anticancer treatment for HCC, including an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody
3. Prior orthotopic liver transplantation
4. Prior abdominal irradiation
5. Any major surgery within the 3 weeks prior to enrolment
6. Hepatic encephalopathy
7. Ascites that is refractory to diuretic therapy
8. Is currently receiving anti-cancer therapy (chemotherapy, radiation therapy, immunotherapy or biologic therapy) or has participated or is participating in a study of an IMP or used an investigational device within 4 weeks of the first dose of IMP
9. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy
10. Known history of active Bacillus Tuberculosis (TB)
11. History of known hypersensitivity to any monoclonal antibody or any of their excipients
12. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
13. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
14. Active infection requiring systemic therapy, with exceptions relating to Hepatitis B and C virus infection
15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating Principal Investigator (PI)
16. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
17. Pregnant or breastfeeding
18. Known history of Human Immunodeficiency Virus (HIV; HIV 1/2 antibodies)
19. Received a live vaccine within 30 days of first dose of IMP administration.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Delay to surgery | Up to Day 92
  number of patients experiencing a surgery delay over 6 weeks or later
ORR after neoadjuvant SBRT+Tislelizumab | One day before resection
  ORR on pre-resection imaging according to the RECIST v1.1/ mRECIST criteria
Pathologic response rate on evaluation of the resected specimen | One month after resection
  pCR (pathological complete response), pPR (pathological partial response), MPR (major pathologic response)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 months after resection
  Safety and tolerability of the sequential SBRT/tislelizumab based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 criteria, including all grade irAEs (Immune-related adverse events) and irAE of grade 3/4.

SECONDARY OUTCOMES:
Disease-free survival disease-free survival (DFS) | From date of resection until the date of first documented progression, assessed up to 3 years
  DFS (disease-free survival) after successful curative resection of tumor
Overall survival | From date of resection until the date of death from any cause, assessed up to 5 years
  OS (overall survival) after successful curative resection of tumor

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhao, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang B, Yue J, Shi X, Cui K, Li L, Zhang C, Sun P, Zhong J, Li Z, Zhao L. Protocol of notable-HCC: a phase Ib study of neoadjuvant tislelizumab with stereotactic body radiotherapy in patients with resectable hepatocellular carcinoma. BMJ Open. 2022 Sep 17;12(9):e060955. doi: 10.1136/bmjopen-2022-060955. PMID 36115673
- [Background] Li M, Yue J, Zhang B, Shi X, Cui K, Liu J, Li Z, Zhao L. Interim report of Notable-HCC: a phase Ⅰb study of neoadjuvant PD-1 with stereotactic body radiotherapy in patients with resectable HCC[J]. Annals of Oncology. VOLUME 34, SUPPLEMENT 2, S598-S599, OCTOBER 2023